CLINICAL TRIAL: NCT03371914
Title: Costs, Efficiency and the Role of Management in HIV Prevention Interventions for Female Sex Workers in Nigeria
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to defunding of USAID project that supported the majority of the sites selected in the randomization.
Sponsor: Instituto Nacional de Salud Publica, Mexico (Other)
Collaborators: Society For Family Health (SFH) (Unknown); National Agency for the Control of AIDS (NACA) (Unknown)
Responsible Party: Principal Investigator, Sergio Bautista Arredondo, Director of Health Economics, Instituto Nacional de Salud Publica, Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: INSaludPublica
Record Dates: First submitted 2017-09-16; First posted 2017-12-13 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: HIV/AIDS
Keywords: costing; behavioral intervention; management
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment: Management + data training (Experimental): The treatment group in the study will receive a 5-day training. The first two days of the training will consist of introducing the data collection tools and collecting baseline data. Days three through five of the training will consist of a variety of management topics.
  On a monthly basis, the treatment group will receive data visualizations that will compare their site's performance that month to pervious performance and to other sites in the study. Both treatment and control groups will collect information regarding input costs and number of services provided on a monthly basis.
  Interventions: Behavioral: Management training and data feedback
- Control: data training only (No Intervention): The control group will receive only a 2-day training which will focus on data collection alone. Both treatment and control groups will collect information regarding input costs and number of services provided on a monthly basis.

INTERVENTIONS:
Behavioral: Management training and data feedback — The management training will consist of a variety of management topics, such as financial, workplace and staff management. The training will include a number of tools that the managers will be expected to bring back with them and use regularly at their site. There will be monthly refresher trainings for the managers via an online platform, where participants will interact about the topics covered in the training and others relevant to their work as managers. Participants will also receive monthly visualizations that compare the data that they enter via tablet monthly to both (1) their baseline data, and (2) to other sites' data. Outcomes that will be measured and reported back to sites include cost per client tested, number of condoms distributed, and number of FSW reached by educational interventions.
  Arms: Treatment: Management + data training

SUMMARY:
This study seeks to measure the costs associated with HIV prevention service delivery to female sex workers (FSW) in Nigeria, as well as examine the relationship between management practices at the community-based organizations (CBOs) and costs. To complete these goals, the study will collect both retrospective and prospective data from CBOs and from centralized information from study partners (Society for Family Health, SFH). In the prospective section of the study, CBOs will be sampled and assigned to either treatment or control groups. Data collected at the CBOs will be aggregated by the CBO managers, and those in the treatment group will receive feedback on their performance on a monthly basis. Those in the treatment group will additionally receive a management training to guide their management practices. Researchers hypothesize that there will be improvements in management indicators and therefore decreases in costs at CBOs in the treatment group. Results will be disseminated to local, national, and international stakeholders.

ELIGIBILITY:
Inclusion Criteria:

* Clusters: community-based organizations that serve female sex workers under Society for Family Health, through the SHIPs or Global Fund grants
* Participants: managers ("officers") that oversee the functions of the organization and supervise volunteer staff

Exclusion Criteria:

* Clusters: excludes organizations not serving female sex workers and not working under Society for Family Health, through Global Fund or SHIPs grants
* Participants: excludes anyone not explicitly working as a manager overseeing volunteer implementation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-08-12 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Change in cost per female sex worker reached by HIV education services | Two years
  This measures the total cost of HIV education provision, divided by the number of female sex workers (FSWs) reached by the service.
Change in cost per female sex worker tested | Two years
  This measures the total cost of HIV testing and counseling, divided by the number of FSWs tested.
Change in cost per female sex worker treated for STIs (sexually transmitted infections) | Two years
  This measures the total cost of STI treatment, divided by the number of FSWs treated for any STI.
Change in cost per female sex worker tested positive | Two years
  This measures the total cost of HIV testing and counseling, divided by the number of FSWs tested positive for HIV.

SECONDARY OUTCOMES:
Productivity of HIV education | Two years
  Productivity of the organizations will be measured as the number of outputs produced for the HIV education intervention-number of FSW reached by HIV education.
Productivity of HIV testing | Two years
  Productivity of the organizations will be measured as the number of outputs produced for the HIV testing and counseling interventions-number of FSW tested for HIV.
Productivity of STI treatment | Two years
  Productivity of the organizations will be measured as the number of outputs produced for the STI treatment intervention-number of FSW treated for STIs.
Job satisfaction | Two years
  Measured through a composite score of five Likert scale questions about satisfaction, answers ranging from 1-5, 1 being "very dissatisfied" and 5 being "very satisfied".

CONTACTS AND LOCATIONS:
Locations (1):
- Society for Family Health, Headquarters, Abuja, Nigeria

REFERENCES:
- [Derived] Bautista-Arredondo S, Nance N, Salas-Ortiz A, Akeju D, Oluwayinka AG, Ezirim I, Anenih J, Chima C, Amanze O, Omoregie G, Ogungbemi K, Aliyu SH. The role of management on costs and efficiency in HIV prevention interventions for female sex workers in Nigeria: a cluster-randomized control trial. Cost Eff Resour Alloc. 2018 Oct 23;16:37. doi: 10.1186/s12962-018-0107-x. eCollection 2018. PMID 30386184